CLINICAL TRIAL: NCT07224568
Title: INTERCEPT-GPC3: Interleukin-15 and -21 Armored Glypican-3 Specific Chimeric Antigen Receptor Expressing Autologous T-cells in Adults With GPC3-positive Solid Tumors
Brief Title: Cytokine Armored GPC3 Specific Chimeric Antigen Receptor Expressing T-cells in Adults With Solid Tumors
Acronym: INTERCEPT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director - Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTERCEPT
Record Dates: First submitted 2025-10-28; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor (Excluding CNS); Hepatocellular Carcinoma; Liver Cell Carcinoma; Liposarcoma; Yolk Sac Tumor; Rhabdomyosarcoma
Keywords: CAR T cell; Adult; Non-CNS Tumor; Liver Cancer; Solid Tumor; GPC3; Glypican
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liposarcoma; Endodermal Sinus Tumor; Rhabdomyosarcoma; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SC-CAR.GPC3xIL15.21 T cells (Experimental): Autologous SC-CAR.GPC3xIL15.21 T cell product infused as a single infusion.
  Interventions: Biological: SC-CAR.GPC3xIL15.21 CAR T cells

INTERVENTIONS:
Biological: SC-CAR.GPC3xIL15.21 CAR T cells — Autologous SC-CAR.GPC3xIL15.21 T cell products infusion

SUMMARY:
This Phase 1, open-label, non-randomized study will enroll adult subjects with relapsed or refractory non-central nervous system (CNS) malignant solid tumors expressing glypican-3 (GPC3) to examine the safety, feasibility, and efficacy of administering T cell products derived from peripheral blood mononuclear cells (PBMC) that have been genetically modified to co-express a GPC3-specific chimeric antigen receptor (CAR), interleukin (IL)-15 and IL-21 as well as the inducible caspase 9 (iC9) suicide gene (SC-CAR.GPC3xIL15.21 T cells).

An adult participant meeting all eligibility criteria and meeting none of the exclusion criteria will have a blood sample collected, which will be used to bioengineer the CAR T cells targeting their tumor.

DETAILED DESCRIPTION:
Study Overview

This study is testing a different treatment which uses the body's own immune system to recognize and kill the cancer cells, called chimeric antigen receptor (CAR) T cells. Some solid tumors express a specific type of molecule called glypican-3 or GPC3. Seattle Children's Therapeutics (SCTx) are able to insert a new gene (a piece of DNA that contains a set of instructions for the body) into T cells which are a type of immune system cell. This is how SCTx make CAR T cells: they will insert a gene that will program the CAR T cell to recognize GPC3 to make GPC3-CAR T cells. To make GPC3-CAR T cells more effective against tumor cells, SCTx also added two genes called IL15 and IL21 which help CAR T cells grow better and stay in the blood longer. The investigators think that this will kill tumors better. When this was done in the laboratory, the investigators found that this mixture of GPC3-CAR, IL15, and IL21 in T cells killed tumor cells better when compared with GPC3-CAR T cells that did not have IL15 and IL21. This research study will use these cells (named GPC3xIL15.21) to treat patients with solid tumors that express GPC3 on their surface. The GPC3xIL15.21 CAR T cells are an investigational product and have not been approved by the Food and Drug Administration.

The investigators also wanted to make sure that we could stop the GPC3xIL15.21 CAR T cells from growing in the blood if there are any bad or severe side effects. To do so, a gene called iCasp9 was inserted into the GPC3xIL15.21 CAR T cells. This the GPC3xIL15.21 CAR T cells in the blood to be eliminated when a medicine called AP1903 (also known as rimiducid) is given. Rimiducid is an experimental medicine that has been tested in humans, with no known bad side effects. This medicine is only intended to be used to get rid of the GPC3xIL15.21 CAR T cells if participants develop dangerous side effects. Approximately 21 people will participate in this study.

Treatment plan

The investigators would first confirm that the participant tumor expresses GPC3. Upon confirmation, a maximum of approximately 6 tablespoons (or 90 mL) of blood will be drawn and sent to SCTx to make the CAR T cells.

After the CAR T cells are made and treatment eligibility has been verified, participants will come to the Fred Hutch Cancer Centre for treatment and close monitoring for about one month. Participants will be given lymphodepleting chemotherapy for 3 days, using cyclophosphamide and fludarabine to make room for the CAR T cells, followed by CAR T cell infusion IV.

This is a dose escalation study, which means that the investigators do not know the highest safe dose of CAR T cells. The dose each patient gets depends on how many participants get the agent before that patient and how they react. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the treatments will be given at Fred Hutch Cancer Centre.

After treatment, participants will be monitored closely for a month to monitor for side effects and response to treatment. After this month, participants would continue to be followed for 15 years after they receive their CAR T cells, with visits becoming less frequent the longer it has been since CAR T cell infusion.

ELIGIBILITY:
1. Procurement Eligibility

   Inclusion Criteria:
   * Diagnosis of a solid tumor expressing GPC3
   * Karnofsky score of >=60%
   * Life expectancy of >16 weeks
   * Informed consent explained to, understood by and signed by participant or participant's legally authorized representative

   For patients with hepatocellular carcinoma only:
   * Barcelona Liver Cancer Stage A, B or C
   * Child-Pugh-Turcotte Score <7

   Exclusion Criteria:
   * History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies.

     * History of organ transplantation
     * Known HIV positivity
     * Active bacterial, fungal, or viral infection (except Hepatitis B or Hepatitis C virus infections)
2. Treatment eligibility

Inclusion Criteria:

* Karnofsky score of >=60%
* Life expectancy of >16 weeks
* Informed consent explained to, understood by and signed by patient/guardian.
* Adequate organ function
* Adequate laboratory values
* Refractory or relapsed disease after treatment with up- front therapy and at least one salvage treatment cycle
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/guardian.

For patients with hepatocellular carcinoma only:

* Barcelona Liver Cancer Stage A, B or C
* Child-Pugh Turcotte Score <7

Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies.

  * History of organ transplantation
  * Known HIV positivity
  * Active bacterial, fungal, or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Pregnancy or lactation
* Systemic steroid treatment (≥ 0.5 mg prednisone equivalent/kg/day, dose adjustment or discontinuation of medication must occur at least 24hrs prior to CAR T cell infusion)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2045-08 (Estimated)

PRIMARY OUTCOMES:
The number of successfully manufactured SC-CAR.GPC3xIL15.21 T cell products will be assessed | 28 days
  The proportion of SC-CAR.GPC3xIL15.21 T cell products that are approved for release after up to 2 grow attempts will be measured.
To determine the safety of escalating doses of an intravenous injection of SC-CAR.GPC3xIL15.21 T cells in adults with relapsed or refractory GPC3-positive solid tumors after lymphodepleting chemotherapy based on frequency of adverse events based on CTCAE | 42 days
  The type, frequency, severity, and duration of adverse events will be tabulated and summarized

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of SC-CAR.GPC3xIL15.21 T cells in treating patients with GPC3-positive solid tumors after lymphodepleting chemotherapy. | 42 days
  The MTD will be estimated based on the type, frequency, severity, and duration of adverse events reported for each subject at the completion of the dose escalation phase.
To assess the response rate in patients with relapsed or refractory GPC3-positive solid tumors infused with SC-CAR.GPC3xIL15.21 T cells. | 42 days
  Response and progression will be evaluated in this study using the international RECIST Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, Study Director — Seattle Children's Hospital; Corinne Summers, Study Director — Seattle Children's Hospital
Locations (1):
- Fred Hutch Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No